CLINICAL TRIAL: NCT03211494
Title: Does Automated Closed-Loop Ventilation Reduce the DRiving Pressure Levels in Patients With ARDS (AiRDRoP) - a Single-Center Crossover Study and Randomized Controlled Trial
Brief Title: Does Automated Closed-Loop Ventilation Reduce the DRiving Pressure Levels in Patients With ARDS
Acronym: AiRDRoP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected low recruitment rate
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AiRDRoP
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: ARDS
Keywords: Mechanical ventilation; Driving pressure; Closed-loop ventilation; Esophageal catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lung protective ventilation (Active Comparator): Use of conventional lung protective ventilation, according to the ARDSnet guidelines
  Interventions: Other: Conventional lung protective ventilation
- INTELLiVENT-ASV (Active Comparator): Use of INTELLiVENT-ASV
  Interventions: Device: INTELLiVENT-ASV

INTERVENTIONS:
Device: INTELLiVENT-ASV — INTELLiVENT-ASV, with software 2.60
  Other Names: automated closed-loop ventilation
  Arms: INTELLiVENT-ASV
Other: Conventional lung protective ventilation — Lung protective ventilation according to the ARDSnet guidelines
  Arms: Conventional lung protective ventilation

SUMMARY:
The objective of this crossover study and randomized controlled trial (RCT) is to compare ΔP levels during INTELLiVENT®-ASV with conventional lung protective ventilation in the acute and sub-acute phase of moderate or severe ARDS.

A total of 48 adult patients admitted to intensive care units with moderate or severe ARDS will be included. In the acute phase patients will receive 4 hours of INTELLiVENT-ASV ventilation and 4 hours of conventional lung protective ventilation in random order. After these two blocks the patients are allocated into either the INTELLiVENT-ASV arm or the conventional lung protective ventilation arm.

in the sub-acute phase patients will be assessed every day until day 7 or extubation, whichever comes first.

Primary endpoint is the transpulmonary transpulmonary (ΔP). Secondary endpoints of both studies include other ventilator settings and ventilation parameters, as well as time spent at a ΔP level of 15 cm H2O or higher.

DETAILED DESCRIPTION:
- Objective:

The objective of this crossover study and randomized controlled trial (RCT) is to compare ΔP levels during INTELLiVENT®- adaptive support ventilation (ASV) with conventional lung protective ventilation in the acute and sub-acute phase of moderate or severe ARDS.

- Study design:

Single center crossover study (in the acute phase) and RCT (in the sub-acute phase).

- Study population:

The study population consists of 48 consecutive intubated and ventilation patients with moderate or severe ARDS according to the Berlin definition with an anticipated duration of mechanical ventilation of > 24 hours.

- Sample size calculation:

The sample size is computed based on the hypothesis that ventilation with INTELLiVENT®-ASV is associated with a reduction in the ΔP level of 5 cm H2O. We based this power calculation on unpublished data from a published cohort of ARDS patients29 and data from an abstract31.

For the RCT, a sample size of 20 patients in each group has 90% statistical power to detect a difference in the ΔP level of 5 cm H2O, with means of 15 and 10 cm H2O, respectively, assuming an effect size (f) of 0.4 using a repeated measures ANOVA with a 0.05 two-sided significance level.

The sample size is increased by 20% to correct for early dropouts (i.e., before day 7) and patients in whom it is impossible to measure the ΔP level, meaning that each group will contain 24 patients. Therefore, the total sample size of this study will be 48 patients.

We expect less variation in the crossover than in the RCT. Next, in this part of the study patients serve as their own control. Therefore, with this sample size we will have sufficient power for the crossover.

- Patient allocation:

Crossover study - Data will be collected during two blocks of four hours; one block of conventional lung protective ventilation, and one block of INTELLiVENT®-ASV. The two blocks will take place in randomized order. Both ventilation strategies are frequently used in our ICU. INTELLiVENT®-ASV is a relatively new ventilatory mode that was successfully implemented in our intensive care unit in 2016, especially in patients with ARDS.

Randomized controlled trial - After the crossover, patients are randomly allocated to conventional lung protective ventilation5, meaning that the ventilator is set to pressure controlled mode, or INTELLiVENT®-ASV.

- Ventilator settings:

Cross-over study

During conventional lung protective ventilation, the attending physician sets the ventilator according to the local ventilation protocol. The fraction of inspired oxygen (FiO2) is adjusted to maintain an oxygen saturation of 92 to 96% and/or a PaO2 of > 8 kPa. The respiratory rate is adjusted to maintain a blood pH of 7.25 to 7.45. The lowest level of positive end-expiratory pressure (PEEP) is 5 cm H2O; allowed PEEP-FiO2 are in concordance with the ARDS network recommendations;5 these combinations are based on two large RCTs in ARDS patients, and is standard practice in our unit.

During INTELLiVENT®-ASV, the attending physician sets the target for et-CO2 to maintain a blood pH of 7.25 to 7.45. The target for oxygen saturation is set at 92- 96%. The lowest level of PEEP is kept at 5 cm H2O.

Of note, INTELLiVENT®-ASV is available on all ventilators used in patients with ARDS. Since both ventilation strategies can be applied with these ventilators, there is no need to disconnect a patient from the ventilator. Also, switching between ventilatory modes is a standard procedure in our ICU. However, for the purpose of this study it is protocolized.

Randomized controlled trial

Settings are similar for the RCT as for the crossover study.

- Statistical analysis:

Primary study parameters

The primary outcome, the (transpulmonary) ΔP level, is analyzed using a repeated measures ANOVA. The effect mediation of ventilator parameters on the (transpulmonary) ΔP is analyzed by mediation analysis. P-values of 0.05 are used for statistical significance. When appropriate, statistical uncertainty will be expressed by the 95% confidence levels. All statistical analysis will be performed with the R language and environment for statistical computing.

Secondary study parameters

Continuous normally distributed variables will be expressed by their mean and standard deviation or when not normally distributed as medians and their interquartile ranges. Categorical variables will be expressed as n (%). To test groups Student's t test will be used, if continuous data is not normally distributed the Mann-Whitney U test will be used. Categorical variables will be compared with the Chi-square test or Fisher's exact tests. Time dependent data will be analyzed using a proportional hazard model adjusted for possible imbalances of patients' baseline characteristics. Analysis will be performed with R statistics version 3.0.2. Patient characteristics will be compared and described by appropriate statistics.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU of the AMC
* Intubated and mechanically ventilated
* Within 24 hours of initial diagnosis of ARDS
* Moderate or severe ARDS (according to the Berlin definition for ARDS)

Exclusion Criteria:

* Age < 18 years
* Patients previously included in this study
* Patients participating in other interventional trials that could influence ventilator settings and ventilation parameters
* Patients with suspected or confirmed pregnancy
* Patients with increased (of > 15 mmHg) or uncontrollable intracranial pressure
* Patients in whom esophageal pressure measurement is contra-indicated (severe bleeding diathesis, suspicion of or known pharyngeal or esophageal obstruction, esophageal ulcers, varices or strictures)
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Transpulmonary driving pressure level | during the course of mechanical ventilation (max. 7 days)
  The driving pressure of the lungs system, difference between end-inspiratory and end-expiratory pressure

SECONDARY OUTCOMES:
Respiratory system driving pressure level | during the course of mechanical ventilation (max. 7 days)
  The driving pressure of the respiratory system, difference between Pplat and PEEP
Tidal volume | during the course of mechanical ventilation (max. 7 days)
  Volume of a breath
PEEP level | during the course of mechanical ventilation (max. 7 days)
  Positive end-expiratory pressure
Pplat level | during the course of mechanical ventilation (max. 7 days)
  Plateau pressure
Ppeak level | during the course of mechanical ventilation (max. 7 days)
  Peak pressure
RRset | during the course of mechanical ventilation (max. 7 days)
  set respiratory rate
RRmeasured | during the course of mechanical ventilation (max. 7 days)
  measured respiratory rate
FiO2 | during the course of mechanical ventilation (max. 7 days)
  Fraction of inspired oxygen
etCO2 | during the course of mechanical ventilation (max. 7 days)
  end tidal carbondioxide
spO2 | during the course of mechanical ventilation (max. 7 days)
  peripheral oxygen saturation
VCO2 | during the course of mechanical ventilation (max. 7 days)
  volume of expired oxygen
PaCO2 | during the course of mechanical ventilation (max. 7 days)
  Partial pressure of arterial carbondioxide
PaO2 | during the course of mechanical ventilation (max. 7 days)
  Partial pressure of arterial oxygen
saO2 | during the course of mechanical ventilation (max. 7 days)
  arterial oxygen saturation
pH | during the course of mechanical ventilation (max. 7 days)
  acidity of the arterial blood
HCO3 | during the course of mechanical ventilation (max. 7 days)
  Bicarbonate
Time spent at high driving pressure | during the course of mechanical ventilation (max. 7 days)
  Time spent at a driving pressure of more than 14 cm H2O

CONTACTS AND LOCATIONS:
Overall Officials: David MP van Meenen, MD, MSc, Study Director — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Marcus J Schultz, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Marcello Gama de Abreu, MD, PhD, Study Chair — Department of Anesthesiology and Intensive Care Medicine, University Hospital Carl Gustav Carus, Technical University Dresden, Germany; Ary Serpa Neto, MD, MSc, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam, The Netherlands; Paolo Pelosi, MD, PhD, Principal Investigator — Department of Surgical Sciences and Integrated Diagnostics, University of Genoa, Italy; Jitske R Rogmans, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Lennard HL Pennekamp, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Frank C Dullemeijer, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Marco Maggiorini, MD, PhD, Principal Investigator — Department of Intensive Care, Universitatsspital, Zurich; Dominik Novotni, MD, PhD, Study Chair — Hamilton Medical AG; Alexandra Gerlach, Principal Investigator — Hamilton Medical AG; Job BM van Woensel, MD, PhD, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Jean-Michel Arnal, MD, PhD, Study Chair — Department of Intensive Care, Intercommunal hospital, Toulon; Patricia Rocco, MD, PhD, Principal Investigator — Laboratory of pulmonary investigation, Federal University, Rio de Janeiro; Dave A Dongelmans, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buiteman-Kruizinga LA, van Meenen DMP, Bos LDJ, van der Heiden PLJ, Paulus F, Schultz MJ. A closed-loop ventilation mode that targets the lowest work and force of breathing reduces the transpulmonary driving pressure in patients with moderate-to-severe ARDS. Intensive Care Med Exp. 2023 Jul 14;11(1):42. doi: 10.1186/s40635-023-00527-1. PMID 37442844